CLINICAL TRIAL: NCT01453985
Title: Full-Thickness-Gastroplication For The Treatment Of Gastroesophageal Reflux Disease GERD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: General Public Hospital Zell am See (Other)
Responsible Party: Sponsor
Other Study IDs: Zell04
Record Dates: First submitted 2011-10-12; First posted 2011-10-18 (Estimated); Last update posted 2011-10-18 (Estimated); Status verified 2011-10

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux

ARMS (1):
- Full-Thickness-Gastroplication (Experimental)
  Interventions: Procedure: Full-Thickness-Gastroplication

INTERVENTIONS:
Procedure: Full-Thickness-Gastroplication

SUMMARY:
This is a prospective study to extensively evaluate subjective patient parameters on quality of life, reflux-symptoms, side effects, medication-use and measurements of esophageal manometry and Impedance-pH-Monitoring after Full-Thickness-Gastroplication.

ELIGIBILITY:
Inclusion Criteria:

* persistent or recurrent symptoms despite continuous medical treatment, at least one typical reflux symptom (heartburn/ regurgitation/dysphagia/epigastric pain) and/or at least one atypical reflux symptom (cough/ asthma/hoarseness/distortion of taste), pathologic esophageal acid exposure as documented by a reflux-related DeMeester score ≥14.7, and symptom correlation ≥50%, and/or reflux episodes >73.

Exclusion Criteria:

* any distinct hiatal hernia detectable by gastroscopy or barium radiography, dysphagia, esophageal strictures, poor physical status (American Society of Anesthesiologists (ASA) scores III and IV) and pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Quality of Life

CONTACTS AND LOCATIONS:
Locations (1):
- General public hospital Zell am See, Zell am See, Austria

REFERENCES:
- [Derived] Koch OO, Kaindlstorfer A, Antoniou SA, Spaun G, Pointner R, Swanstrom LL. Subjective and objective data on esophageal manometry and impedance pH monitoring 1 year after endoscopic full-thickness plication for the treatment of GERD by using multiple plication implants. Gastrointest Endosc. 2013 Jan;77(1):7-14. doi: 10.1016/j.gie.2012.07.033. Epub 2012 Sep 26. PMID 23021166